CLINICAL TRIAL: NCT07287644
Title: A Phase 2, Dose Ranging, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of BFB759 in Patients With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study Evaluating BFB759 in Moderate to Severe Hidradenitis Suppurativa
Acronym: COMPASS 2-HS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bluefin Biomedicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-BFB759-003; COMPASS 2-HS (Other: Sponsor)
Record Dates: First submitted 2025-11-13; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; acne inversa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active - high dose (Experimental): BFB759 loading dose followed by BFB759 maintenance high dose every 2 weeks (Q2W) through Week 14 (inclusive), which is followed by placebo Q2W at Weeks 16 through 30 (inclusive).
  Interventions: Biological: BFB759
- Active - low dose (Experimental): BFB759 loading dose followed by BFB759 maintenance mid-dose Q2W through Week 14 (inclusive).
  Interventions: Biological: BFB759
- Placebo (Placebo Comparator): Placebo Q2W for 14 weeks. At Week 16, participants in Placebo group who are still enrolled in the study and receiving treatment will be re-randomized (1:1) into 2 groups (Cross 1 and Cross 2) to receive BFB759
  * Cross 1 will receive BFB759 loading dose followed by BFB759 maintenance low-dose Q2W through Week 30 (inclusive).
  * Cross 2 will receive BFB759 loading dose followed by BFB759 maintenance mid-dose Q2W through Week 30 (inclusive).
  Interventions: Other: Placebo for BFB759

INTERVENTIONS:
Biological: BFB759 — BFB759 is a human mAb that inhibits multiple pro-inflammatory cytokines that contribute to the pathogenesis of multiple disease processes characterized by aberrant inflammation, including hidradenitis suppurativa.
  Arms: Active - high dose; Active - low dose
Other: Placebo for BFB759 — Placebo for BFB759
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled study where subjects are participating for approximately 36 to 40 weeks. The study compares how well BFB759 works and how safe it is compared with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Are adults (18 to 75 years) with a diagnosis of hidradenitis suppurativa for at least one year.
* Have moderate to severe disease not well controlled by systemic antibiotic treatment.
* Are willing to follow study instructions, attend regular visits, and avoid certain other medications during the study.

Exclusion Criteria:

* Have certain infections or other immune conditions.
* Recently used medications that could interfere with the study.
* Are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of BFB759 in HS | Baseline to Week 16 and baseline to Week 32
  To evaluate the efficacy of BFB759 in adult male and female participants with HS as measured by the change in the number of abscesses and inflammatory nodules (AN count).

SECONDARY OUTCOMES:
Evaluate the clinical activity of BFB759 using HiSCR50 | Baseline to Week 16 and baseline to Week 32
  The HiSCR50 is defined as at least a 50% reduction in inflammatory lesion count [the sum of Abscesses and Inflammatory Nodules (AN)] and no increase in abscess count and no increase in draining fistula count relative to baseline. The threshold of 50% reduction in AN count is the defined level that is clinically appropriate and meaningful to the patient regarding improvement in quality of life and pain level.
Evaluate the safety/tolerability of BFB759 | routinely over 21 months (about 22 visits during the course of study)
  Record how well participants tolerate the treatment over time by recording the incidence and severity of treatment-emergent adverse events (as described by CTCAE Version 5.0)
To evaluate the clinical activity of BFB759 using the International Hidradenitis Suppurativa Severity Score System (IHS4) | Baseline to Week 16 and baseline to Week 32
  The IHS4 is a validated tool to dynamically assess HS severity that can be used both in real-life and the clinical trials setting (Zouboulis, 2017). It is calculated by counting nodules, abscesses and dTs/sinus tracts, and calculating a total score. IHS4 = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of dTs multiplied by 4].
To evaluate the clinical activity of BFB759 using the Skin Pain Numerical Rating Scale (NRS) | Baseline to Week 16 and baseline to Week 32
  The Skin Pain NRS is a single self-reported item designed to measure skin pain severity over the previous 24 hours. The following question is asked, and the response is marked on an 11 point scale where 0 equals no pain and 10 equals the worst pain imaginable.
To evaluate the clinical activity of BFB759 using the Hidradenitis Suppurativa-Investigator Global Assessment (HS-IGA) | Baseline to Week 16 and baseline to Week 32
  The HS IGA is a HS-specific global assessment. It is a 6 point ordinal scale based on objective lesion counts (Garg, 2022). Scores are calculated by the sum of abscesses, nodules (inflammatory or noninflammatory) and tunnels (draining or nondraining) in either the upper body regions or the lower body regions, whichever is greater. Scores are assigned as follows: 0 (0 1 lesions), 1 (2 5 lesions), 2 (6 10 lesions), 3 (11 15 lesions), 4 (16 20 lesions), and 5 (>20 lesions).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Skin Care Research, Boca Raton, Florida
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Clinical Trials Management, LLC, Tampa, Florida
  - Clinical Trials Management, LLC, Metairie, Louisiana

IPD SHARING:
Plan to Share IPD: No